CLINICAL TRIAL: NCT04581629
Title: A Phase 2b, Open-label Dose-ranging Study Evaluating the Safety, Tolerability, Pharmacodynamics and Pharmacokinetics, and Efficacy of CLTX-305 (Encaleret) in Autosomal Dominant Hypocalcemia (ADH) Type 1
Brief Title: Safety, Tolerability, and Efficacy of Encaleret in Participants With Autosomal Dominant Hypocalcemia (ADH) Type 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Calcilytix Therapeutics, Inc., a BridgeBio company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CLTX-305-201
Record Dates: First submitted 2020-09-16; First posted 2020-10-09 (Actual); Results first posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-10

CONDITIONS: Autosomal Dominant Hypocalcemia (ADH); Autosomal Dominant Hypocalcemia Type 1 (ADH1)
MeSH Terms: conditions — Hypercalciuric Hypocalcemia, Familial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Ascending + Steady-State Dose (Experimental): Period 1: Participants will receive an ascending dose of encaleret once daily for the first 3 days. Participants will then receive an individualized dose of encaleret twice daily for 2 days.
  Period 2: Participants will receive encaleret twice daily for 5 days at a single dose level based on responses from Period 1.
  Period 3: After completion of Period 2, participants will be eligible to receive encaleret for an additional 24 weeks.
  Long-Term Extension (LTE): At the end of the study, participants will also have an option to receive encaleret for up to an additional 2 years.
  Interventions: Drug: Encaleret
- Cohort 2: Steady-State Dose (Experimental): Participants will directly be enrolled into Period 2, and receive encaleret twice daily at a dose based on data and responses from Cohort 1 Period 1.
  Period 2: Participants will receive encaleret twice daily for 5 days.
  Period 3: After completion of Period 2, participants will be eligible to receive encaleret for an additional 24 weeks.
  LTE: At the end of the study, participants will also have an option to receive encaleret for up to an additional 2 years.
  Interventions: Drug: Encaleret

INTERVENTIONS:
Drug: Encaleret — Tablets administered orally
  Other Names: CLTX-305

SUMMARY:
The primary purpose of this study is to evaluate the safety, tolerability and effectiveness of encaleret in participants with Autosomal Dominant Hypocalcemia Type 1 (ADH1).

ELIGIBILITY:
Key Inclusion Criteria:

* Be able to understand and sign a written informed consent or assent form, which must be obtained prior to initiation of study procedures.
* Postmenopausal women are allowed to participate in this study
* Body mass index (BMI) ≥ 18.5 to < 39 kilograms (kg)/square meter (m^2)
* Have an activating mutation of the Calcium-sensing receptor (CASR) gene
* Participants being treated with thiazide diuretics may be enrolled if they are willing and able to discontinue thiazides
* Participants being treated with strong Cytochrome P3A4 (CYP3A4) inhibitors should ideally, if clinically appropriate, discontinue these medications during the screening period
* Participants being treated with magnesium or potassium citrate supplements should discontinue such treatment starting on Day -1 during Period 1 and Period 2 and may be asked to discontinue treatment during Period 3

Key Exclusion Criteria:

* History of treatment with parathyroid hormone (PTH) 1-84 or 1-34 within the previous 3 months
* History of hypocalcemic seizure within the past 3 months
* Blood 25-OH Vitamin D level < 25 nanograms (ng)/milliliter (mL)
* Participants with hemoglobin (Hgb) < 13 grams (g)/deciliter (dL) for men and < 12 g/dL for women
* Estimated glomerular filtration rate (eGFR) < 25 mL/minute/1.73 m^2 using Chronic Kidney Disease Epidemiology Collaboration (for participants <18 years old the Schwartz equation will be calculated)
* 12-lead resting electrocardiogram (ECG) with clinically significant abnormalities
* Participants with positive hepatitis B surface antigen (HBsAg), hepatitis A immunoglobulin M (IgM), or human immunodeficiency virus (HIV) viral serology test results at the Screening Visit
* Pregnant or nursing (lactating) women
* History of drug or alcohol dependency within 12 months preceding the Screening Visit
* History of thyroid or parathyroid surgery
* Current participation in other investigational drug studies
* Unwillingness to refrain from blood donation within 12 weeks prior to Screening Visit from the start of the study enrollment through one year after the last dose of the study drug

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-09-20 (Actual); Primary Completion 2023-09-07 (Actual); Study Completion 2023-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Calcilytix Medical Director, Study Director — Calcilytix Therapeutics, Inc., a BridgeBio company
Locations (1):
- National Institutes of Health (NIH) Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 13 participants were enrolled. Participants were enrolled in 3 periods sequentially to receive encaleret, Period 1(inpatient), Period 2(inpatient), and Period 3(outpatient). 6 participants were enrolled into Period 1. Participants who completed Period 1 enrolled into Period 2, and 7 additional participants enrolled into Period 2. 13 participants who completed Period 2 enrolled into Period 3. As pre-specified, data were collected and reported pooled for Period 1, 2 and 3 respectively.
Groups:
- Period 1: Encaleret: In Period 1 (5 days), participants received an ascending dose of oral encaleret once daily (QD) for the first 3 days (Day 1: 30 mg QD, Day 2: 10, 60 or 90 mg QD, Day 3: 20, 40, 60, 90, 120 or 180 mg QD). Participants then received an individualized dose of oral encaleret twice daily (BID) for 2 days (Day 4 and Day 5: 10 to 180 mg BID).
- Period 2: Encaleret: In Period 2 (5 days), participants received encaleret BID for 5 days at dose levels based on responses from Period 1. On Day 1 and Day 2, participants received 10 to 240 mg BID. On Day 3 to Day 5, participants received 10 to 360 mg BID.
- Period 3: Encaleret: In Period 3 (24 weeks), participants received encaleret for an additional 24 weeks. Participants received encaleret at an initial dose based on tolerance and response to the encaleret dose at the end of Period 2.
Period: Period 1 (5 Days)
Arm/Group | Period 1: Encaleret | Period 2: Encaleret | Period 3: Encaleret
Started | 6 | 0 (This group did not enroll participants for Period 1.) | 0 (This group did not enroll participants for Period 1.)
Received at Least One Dose of Study Treatment | 6 | 0 (This group did not enroll participants for Period 1.) | 0 (This group did not enroll participants for Period 1.)
Completed | 6 | 0 (This group did not enroll participants for Period 1.) | 0 (This group did not enroll participants for Period 1.)
Not Completed | 0 | 0 | 0
Period: Period 2 (5 Days)
Arm/Group | Period 1: Encaleret | Period 2: Encaleret | Period 3: Encaleret
Started | 0 (This group did not enroll participants for Period 2.) | 13 (The 6 participants who completed Period 1 enrolled into Period 2 and 7 additional participants were enrolled into Period 2.) | 0 (This group did not enroll participants for Period 2.)
Received at Least One Dose of Study Treatment | 0 (This group did not enroll participants for Period 2.) | 13 | 0 (This group did not enroll participants for Period 2.)
Completed | 0 (This group did not enroll participants for Period 2.) | 13 | 0 (This group did not enroll participants for Period 2.)
Not Completed | 0 | 0 | 0
Period: Period 3 (24 Weeks)
Arm/Group | Period 1: Encaleret | Period 2: Encaleret | Period 3: Encaleret
Started | 0 (This group did not enroll participants for Period 3.) | 0 (This group did not enroll participants for Period 3.) | 13
Received at Least One Dose of Study Treatment | 0 (This group did not enroll participants for Period 3.) | 0 (This group did not enroll participants for Period 3.) | 13
Completed | 0 (This group did not enroll participants for Period 3.) | 0 (This group did not enroll participants for Period 3.) | 13
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who received at least one dose of study drug in the considered period. As pre-specified, data were collected and are reported pooled for Period 1 and for Periods 2 and 3 combined.
Groups:
- Encaleret: In Period 1 (5 days), participants received an ascending dose of oral encaleret once daily (QD) for the first 3 days (Day 1: 30 mg QD, Day 2: 10, 60 or 90 mg QD, Day 3: 20, 40, 60, 90, 120 or 180 mg QD). Participants then received an individualized dose of oral encaleret twice daily (BID) for 2 days (Day 4 and Day 5: 10 to 180 mg BID).
  In Period 2 (5 days), participants received encaleret BID for 5 days at dose levels based on responses from Period 1. On Day 1 and Day 2, participants received 10 to 240 mg BID. On Day 3 to Day 5, participants received 10 to 360 mg BID.
  In Period 3 (24 weeks), participants received encaleret for an additional 24 weeks. Participants received encaleret at an initial dose based on tolerance and response to the encaleret dose at the end of Period 2.
Arm/Group | Encaleret
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data are reported separately for each period of the study. As pre-specified, data for Periods 2 and 3 are combined as the same participants flowed from Period 2 to Period 3.
  years
    Period 1: number analyzed (Participants) | 6
    Period 1 | 40.0 (17.65)
    Periods 2 and 3 | 38.9 (14.90)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data are reported separately for each period of the study. As pre-specified, data for Periods 2 and 3 are combined as the same participants flowed from Period 2 to Period 3.
  Participants
    Period 1: number analyzed (Participants) | 6
    Period 1: Female | 3
    Period 1: Male | 3
    Periods 2 and 3: Female | 8
    Periods 2 and 3: Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data are reported separately for each period of the study. As pre-specified, data for Periods 2 and 3 are combined as the same participants flowed from Period 2 to Period 3.
  Participants
    Period 1: number analyzed (Participants) | 6
    Period 1: Hispanic or Latino | 0
    Period 1: Not Hispanic or Latino | 6
    Period 1: Unknown or Not Reported | 0
    Periods 2 and 3: Hispanic or Latino | 0
    Periods 2 and 3: Not Hispanic or Latino | 13
    Periods 2 and 3: Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data are reported separately for each period of the study. As pre-specified, data for Periods 2 and 3 are combined as the same participants flowed from Period 2 to Period 3.
  Participants
    Period 1: number analyzed (Participants) | 6
    Period 1: American Indian or Alaska Native | 0
    Period 1: Asian | 0
    Period 1: Native Hawaiian or Other Pacific Islander | 0
    Period 1: Black or African American | 0
    Period 1: White | 6
    Period 1: More than one race | 0
    Period 1: Unknown or Not Reported | 0
    Periods 2 and 3: American Indian or Alaska Native | 0
    Periods 2 and 3: Asian | 0
    Periods 2 and 3: Native Hawaiian or Other Pacific Islander | 0
    Periods 2 and 3: Black or African American | 0
    Periods 2 and 3: White | 13
    Periods 2 and 3: More than one race | 0
    Periods 2 and 3: Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Periods 1, 2 and 3: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Adverse events (AEs) were defined as any untoward medical occurrence associated with the use of an intervention in humans, whether or not considered intervention-related. Treatment-emergence was defined as any AE(s) regardless of relationship to investigational medicinal product (IMP), that had an onset or worsened in severity on or after the first dose of IMP.
Time Frame: Day 1 up to 16 months
Population: Safety Analysis Set included all participants who received at least one dose of study drug in the considered period. As pre-specified in the protocol, data were collected and are presented pooled for Periods 2 and 3.
Measure: Count of Participants; unit: Participants
Groups:
- Periods 2 and 3: Encaleret: In Period 2 (5 days), participants received encaleret BID for 5 days at dose levels based on responses from Period 1. On Day 1 and Day 2, participants received 10 to 240 mg BID. On Day 3 to Day 5, participants received 10 to 360 mg BID.
  In Period 3 (24 weeks), participants received encaleret for an additional 24 weeks. Participants received encaleret at an initial dose based on tolerance and response to the encaleret dose at the end of Period 2.
Arm/Group | Period 1: Encaleret | Periods 2 and 3: Encaleret
Number analyzed (Participants) | 6 | 13
Participants | 5 | 13

2. Primary Outcome: Period 3: Change From Baseline in Albumin-Corrected Blood Calcium Concentrations (cCa)
Time Frame: Baseline, Week 24
Population: Safety Analysis Set included all participants who received at least one dose of study drug in the considered period. As pre-specified in the protocol, data are presented for Period 3 only. As pre-specified, data were collected and are reported pooled for all dose levels in Period 3 and are presented at the specified timepoint.
Measure: Mean (Standard Deviation); unit: milligrams (mg)/deciliter (dL)
Arm/Group | Period 3: Encaleret
Number analyzed (Participants) | 13
milligrams (mg)/deciliter (dL) | 1.9 (0.48)

3. Primary Outcome: Period 3: Rate of Urinary Calcium Excretion
Time Frame: Week 24
Population: Safety Analysis Set included all participants who received at least one dose of study drug in the considered period. As pre-specified in the protocol, data are presented for Period 3 only. Number analyzed = number of participants evaluable at the specified timepoint. As pre-specified, data were collected and are reported pooled for all dose levels in Period 3 and are presented at the specified timepoint.
Measure: Mean (Standard Deviation); unit: mg/24hour (hr)
Arm/Group | Period 3: Encaleret
Number analyzed (Participants) | 13
mg/24hour (hr) | 202 (83)

4. Secondary Outcome: Periods 1 and 2: Intact Parathyroid Hormone (iPTH) Concentrations in the Blood
Description: Blood samples were taken for analysis of iPTH concentrations. iPTH concentrations were analyzed via an electrochemiluminescence immunoassay.
Time Frame: 15 minutes pre-dose on Day 5 of Periods 1 and 2 (Periods were 5 days)
Population: Safety Analysis Set, all participants who received at least 1 dose of study drug in the considered period. As pre-specified in the protocol, data are presented for Periods 1 and 2 only. Overall number of participants analyzed=those evaluable for this endpoint. Number analyzed=those evaluable at specified timepoints. As pre-specified, data were collected and reported pooled for all dose levels in Period 2 at the specified timepoint and per dose at the specified timepoint in Period 1.
Measure: Mean (Standard Deviation); unit: Picograms (pg)/milliliter (mL)
Arm/Group | Period 1: Encaleret | Period 2: Encaleret
Number analyzed (Participants) | 6 | 12
Picograms (pg)/milliliter (mL)
  Period 1: Day 5 (180 mg): number analyzed (Participants) | 6 | 0
  Period 1: Day 5 (180 mg) | 43.8 (34.06) |
  Period 2: Day 5: number analyzed (Participants) | 0 | 12
  Period 2: Day 5 |  | 20.6 (15.87)

5. Secondary Outcome: Periods 1 and 2: Area Under the Concentration-Time Curve Extrapolated to Infinity (AUC0-inf) of Encaleret
Time Frame: Periods 1 and 2: Day 5 (Periods were 5 days)
Population: Pharmacokinetic (PK) Analysis Set included all participants who received at least one dose of study drug and who had at least one non-missing PK concentration result. Overall number of participants analyzed = participants evaluable for this endpoint. Number analyzed = participants evaluable for this endpoint at the specified timepoints. As pre-specified in the protocol, data are presented for Periods 1 and 2 only.
Measure: Mean (Standard Deviation); unit: hour (hr)*nanogram (ng)/milliliter (mL)
Arm/Group | Period 1: Encaleret | Period 2: Encaleret
Number analyzed (Participants) | 6 | 1
hour (hr)*nanogram (ng)/milliliter (mL)
  Period 1: Day 5 AM 180mg: number analyzed (Participants) | 4 | 0
  Period 1: Day 5 AM 180mg | 11283.7 (3556.12) |
  Period 1: Day 5 PM 180 mg: number analyzed (Participants) | 3 | 0
  Period 1: Day 5 PM 180 mg | 13127.7 (2992.61) |
  Period 1: Day 5 PM 120 mg: number analyzed (Participants) | 1 | 0
  Period 1: Day 5 PM 120 mg | 12417.0 (NA) — Standard deviation could not be calculated as there was only 1 participant with evaluable data. |
  Period 2: Day 5 PM 10mg: number analyzed (Participants) | 0 | 1
  Period 2: Day 5 PM 10mg |  | 623.7 (NA) — Standard deviation could not be calculated as there was only 1 participant with evaluable data.

6. Secondary Outcome: Periods 1, 2 and 3: Maximum Plasma Concentration (Cmax) of Encaleret
Time Frame: Periods 1 and 2: Day 5, Period 3: Week 24 (Period was 5 days for Periods 1 and 2; 24 weeks for Period 3)
Population: Pharmacokinetic (PK) Analysis Set included all participants who received at least one dose of study drug and who had at least one non-missing PK concentration result. Overall number of participants analyzed = participants evaluable for the endpoint. Number analyzed = participants evaluable for the endpoint at the specified timepoints. As pre-specified in the protocol, data for Periods 2 and 3 are reported per dose received.
Measure: Mean (Standard Deviation); unit: nanograms (ng)/milliliter (mL)
Arm/Group | Period 1: Encaleret | Period 2: Encaleret | Period 3: Encaleret
Number analyzed (Participants) | 6 | 3 | 2
nanograms (ng)/milliliter (mL)
  Period 1: Day 5 AM 180mg: number analyzed (Participants) | 6 | 0 | 0
  Period 1: Day 5 AM 180mg | 2593.3 (655.89) |  |
  Period 1: Day 5 PM 180 mg: number analyzed (Participants) | 5 | 0 | 0
  Period 1: Day 5 PM 180 mg | 1834.0 (470.46) |  |
  Period 1: Day 5 PM 120 mg: number analyzed (Participants) | 1 | 0 | 0
  Period 1: Day 5 PM 120 mg | 1890.0 (NA) — Standard deviation could not be calculated as there was only 1 participant with evaluable data. |  |
  Period 2: Day 5AM 10 mg: number analyzed (Participants) | 0 | 1 | 0
  Period 2: Day 5AM 10 mg |  | 102.0 (NA) — Standard deviation could not be calculated as there was only 1 participant with evaluable data. |
  Period 2: Day 5AM 30 mg: number analyzed (Participants) | 0 | 3 | 0
  Period 2: Day 5AM 30 mg |  | 223.6 (169.94) |
  Period 2: Day 5AM 60 mg: number analyzed (Participants) | 0 | 1 | 0
  Period 2: Day 5AM 60 mg |  | 496.0 (NA) — Standard deviation could not be calculated as there was only 1 participant with evaluable data. |
  Period 2: Day 5AM 90 mg: number analyzed (Participants) | 0 | 3 | 0
  Period 2: Day 5AM 90 mg |  | 1041.0 (303.40) |
  Period 2: Day 5AM 120 mg: number analyzed (Participants) | 0 | 1 | 0
  Period 2: Day 5AM 120 mg |  | 1720.0 (NA) — Standard deviation could not be calculated as there was only 1 participant with evaluable data. |
  Period 2: Day 5AM 150 mg: number analyzed (Participants) | 0 | 1 | 0
  Period 2: Day 5AM 150 mg |  | 1560.0 (NA) — Standard deviation could not be calculated as there was only 1 participant with evaluable data. |
  Period 2: Day 5AM 180 mg: number analyzed (Participants) | 0 | 3 | 0
  Period 2: Day 5AM 180 mg |  | 1956.7 (748.09) |
  Period 2: Day 5PM 10 mg: number analyzed (Participants) | 0 | 3 | 0
  Period 2: Day 5PM 10 mg |  | 134.3 (34.53) |
  Period 2: Day 5PM 30 mg: number analyzed (Participants) | 0 | 1 | 0
  Period 2: Day 5PM 30 mg |  | 226.0 (NA) — Standard deviation could not be calculated as there was only 1 participant with evaluable data. |
  Period 2: Day 5PM 60 mg: number analyzed (Participants) | 0 | 1 | 0
  Period 2: Day 5PM 60 mg |  | 373.0 (NA) — Standard deviation could not be calculated as there was only 1 participant with evaluable data. |
  Period 2: Day 5PM 90 mg: number analyzed (Participants) | 0 | 3 | 0
  Period 2: Day 5PM 90 mg |  | 822.3 (73.93) |
  Period 2: Day 5PM 120 mg: number analyzed (Participants) | 0 | 1 | 0
  Period 2: Day 5PM 120 mg |  | 1670.0 (NA) — Standard deviation could not be calculated as there was only 1 participant with evaluable data. |
  Period 2: Day 5PM 150 mg: number analyzed (Participants) | 0 | 1 | 0
  Period 2: Day 5PM 150 mg |  | 1590.0 (NA) — Standard deviation could not be calculated as there was only 1 participant with evaluable data. |
  Period 2: Day 5PM 180 mg: number analyzed (Participants) | 0 | 3 | 0
  Period 2: Day 5PM 180 mg |  | 2203.3 (254.23) |
  Period 3: Week 24 5 mg: number analyzed (Participants) | 0 | 0 | 1
  Period 3: Week 24 5 mg |  |  | 44.4 (NA) — Standard deviation could not be calculated as there was only 1 participant with evaluable data.
  Period 3: Week 24 10 mg: number analyzed (Participants) | 0 | 0 | 1
  Period 3: Week 24 10 mg |  |  | 58.6 (NA) — Standard deviation could not be calculated as there was only 1 participant with evaluable data.
  Period 3: Week 24 20 mg: number analyzed (Participants) | 0 | 0 | 2
  Period 3: Week 24 20 mg |  |  | 200.5 (50.20)
  Period 3: Week 24 30 mg: number analyzed (Participants) | 0 | 0 | 1
  Period 3: Week 24 30 mg |  |  | 466.0 (NA) — Standard deviation could not be calculated as there was only 1 participant with evaluable data.
  Period 3: Week 24 60 mg: number analyzed (Participants) | 0 | 0 | 1
  Period 3: Week 24 60 mg |  |  | 403.0 (NA) — Standard deviation could not be calculated as there was only 1 participant with evaluable data.
  Period 3: Week 24 70 mg: number analyzed (Participants) | 0 | 0 | 1
  Period 3: Week 24 70 mg |  |  | 472.0 (NA) — Standard deviation could not be calculated as there was only 1 participant with evaluable data.
  Period 3: Week 24 80 mg: number analyzed (Participants) | 0 | 0 | 1
  Period 3: Week 24 80 mg |  |  | 872.0 (NA) — Standard deviation could not be calculated as there was only 1 participant with evaluable data.
  Period 3: Week 24 120 mg: number analyzed (Participants) | 0 | 0 | 1
  Period 3: Week 24 120 mg |  |  | 1090.0 (NA) — Standard deviation could not be calculated as there was only 1 participant with evaluable data.
  Period 3: Week 24 150 mg: number analyzed (Participants) | 0 | 0 | 1
  Period 3: Week 24 150 mg |  |  | 1110.0 (NA) — Standard deviation could not be calculated as there was only 1 participant with evaluable data.
  Period 3: Week 24 180 mg: number analyzed (Participants) | 0 | 0 | 2
  Period 3: Week 24 180 mg |  |  | 2125.0 (21.21)
  Period 3: Week 24 190 mg: number analyzed (Participants) | 0 | 0 | 1
  Period 3: Week 24 190 mg |  |  | 2080.0 (NA) — Standard deviation could not be calculated as there was only 1 participant with evaluable data.

7. Secondary Outcome: Periods 1, 2 and 3: Time to Maximum Plasma Concentration (Tmax) of Encaleret
Time Frame: Periods 1 and 2: Day 5; Period 3: Week 24 (Period was 5 days for Periods 1 and 2; 24 weeks for Period 3)
Population: as for outcome 6
Measure: Median (Full Range); unit: hour
Arm/Group | Period 1: Encaleret | Period 2: Encaleret | Period 3: Encaleret
Number analyzed (Participants) | 6 | 3 | 2
hour
  Period 1: Day 5 AM 180mg: number analyzed (Participants) | 6 | 0 | 0
  Period 1: Day 5 AM 180mg | 1.1 [1.0 to 3.0] |  |
  Period 1: Day 5 PM 180 mg: number analyzed (Participants) | 5 | 0 | 0
  Period 1: Day 5 PM 180 mg | 1.5 [1.5 to 3.0] |  |
  Period 1: Day 5 PM 120 mg: number analyzed (Participants) | 1 | 0 | 0
  Period 1: Day 5 PM 120 mg | 2.0 [2.0 to 2.0] |  |
  Period 2: Day 5AM 10 mg: number analyzed (Participants) | 0 | 1 | 0
  Period 2: Day 5AM 10 mg |  | 1.5 [1.5 to 1.5] |
  Period 2: Day 5AM 30 mg: number analyzed (Participants) | 0 | 3 | 0
  Period 2: Day 5AM 30 mg |  | 4.0 [1.5 to 4.0] |
  Period 2: Day 5AM 60 mg: number analyzed (Participants) | 0 | 1 | 0
  Period 2: Day 5AM 60 mg |  | 1.5 [1.5 to 1.5] |
  Period 2: Day 5AM 90 mg: number analyzed (Participants) | 0 | 3 | 0
  Period 2: Day 5AM 90 mg |  | 1.5 [1.5 to 4.0] |
  Period 2: Day 5AM 120 mg: number analyzed (Participants) | 0 | 1 | 0
  Period 2: Day 5AM 120 mg |  | 1.5 [1.5 to 1.5] |
  Period 2: Day 5AM 150 mg: number analyzed (Participants) | 0 | 1 | 0
  Period 2: Day 5AM 150 mg |  | 1.5 [1.5 to 1.5] |
  Period 2: Day 5AM 180 mg: number analyzed (Participants) | 0 | 3 | 0
  Period 2: Day 5AM 180 mg |  | 1.5 [1.5 to 4.0] |
  Period 2: Day 5PM 10 mg: number analyzed (Participants) | 0 | 3 | 0
  Period 2: Day 5PM 10 mg |  | 1.4 [0.5 to 1.5] |
  Period 2: Day 5PM 30 mg: number analyzed (Participants) | 0 | 1 | 0
  Period 2: Day 5PM 30 mg |  | 1.5 [1.5 to 1.5] |
  Period 2: Day 5PM 60 mg: number analyzed (Participants) | 0 | 1 | 0
  Period 2: Day 5PM 60 mg |  | 1.5 [1.5 to 1.5] |
  Period 2: Day 5PM 90 mg: number analyzed (Participants) | 0 | 3 | 0
  Period 2: Day 5PM 90 mg |  | 1.5 [0.5 to 1.5] |
  Period 2: Day 5PM 120 mg: number analyzed (Participants) | 0 | 1 | 0
  Period 2: Day 5PM 120 mg |  | 1.5 [1.5 to 1.5] |
  Period 2: Day 5PM 150 mg: number analyzed (Participants) | 0 | 1 | 0
  Period 2: Day 5PM 150 mg |  | 1.5 [1.5 to 1.5] |
  Period 2: Day 5PM 180 mg: number analyzed (Participants) | 0 | 3 | 0
  Period 2: Day 5PM 180 mg |  | 1.5 [1.5 to 1.5] |
  Period 3: Week 24 5 mg: number analyzed (Participants) | 0 | 0 | 1
  Period 3: Week 24 5 mg |  |  | 2.0 [2.0 to 2.0]
  Period 3: Week 24 10 mg: number analyzed (Participants) | 0 | 0 | 1
  Period 3: Week 24 10 mg |  |  | 2.0 [2.0 to 2.0]
  Period 3: Week 24 20 mg: number analyzed (Participants) | 0 | 0 | 2
  Period 3: Week 24 20 mg |  |  | 2.0 [2.0 to 2.0]
  Period 3: Week 24 30 mg: number analyzed (Participants) | 0 | 0 | 1
  Period 3: Week 24 30 mg |  |  | 0.5 [0.5 to 0.5]
  Period 3: Week 24 60 mg: number analyzed (Participants) | 0 | 0 | 1
  Period 3: Week 24 60 mg |  |  | 2.0 [2.0 to 2.0]
  Period 3: Week 24 70 mg: number analyzed (Participants) | 0 | 0 | 1
  Period 3: Week 24 70 mg |  |  | 4.0 [4.0 to 4.0]
  Period 3: Week 24 80 mg: number analyzed (Participants) | 0 | 0 | 1
  Period 3: Week 24 80 mg |  |  | 0.5 [0.5 to 0.5]
  Period 3: Week 24 120 mg: number analyzed (Participants) | 0 | 0 | 1
  Period 3: Week 24 120 mg |  |  | 2.0 [2.0 to 2.0]
  Period 3: Week 24 150 mg: number analyzed (Participants) | 0 | 0 | 1
  Period 3: Week 24 150 mg |  |  | 4.0 [4.0 to 4.0]
  Period 3: Week 24 180 mg: number analyzed (Participants) | 0 | 0 | 2
  Period 3: Week 24 180 mg |  |  | 2.0 [2.0 to 2.1]
  Period 3: Week 24 190 mg: number analyzed (Participants) | 0 | 0 | 1
  Period 3: Week 24 190 mg |  |  | 2.0 [2.0 to 2.0]

8. Secondary Outcome: Periods 2 and 3: Change From Baseline in Blood Calcium Concentration (cCa)
Description: Data values presented are for the change from baseline for the average values at the specified timepoints/visits.
Time Frame: Period 2: Baseline, Day 5 (Period was 5 days), Period 3: Baseline, Week 24 (Period was 24 weeks)
Population: Safety Analysis Set included all participants who received at least one dose of study drug in the considered period. As pre-specified in the protocol, data are presented for Periods 2 and 3 only. Number analyzed = participants evaluable for the endpoint at the specified timepoints. As pre-specified, data were collected and are reported pooled for all dose levels in Period 2 and Period 3 and are presented at the specified timepoints.
Measure: Mean (Standard Deviation); unit: milligram (mg)/ deciliter (dL)
Arm/Group | Period 2: Encaleret | Period 3: Encaleret
Number analyzed (Participants) | 13 | 13
milligram (mg)/ deciliter (dL)
  Period 2: Day 5: number analyzed (Participants) | 13 | 0
  Period 2: Day 5 | 1.5 (0.60) |
  Period 3: Week 24: number analyzed (Participants) | 0 | 13
  Period 3: Week 24 |  | 1.9 (0.48)

9. Secondary Outcome: Period 3: Urinary Calcium Clearance as Assessed by Fractional Excretion
Description: Fractional Excretion of Calcium was derived as (Urine Calcium at the interval considered * Serum Creatinine at the end of the interval considered)/(Serum Calcium at the end of the interval considered * Urine Creatinine at the interval considered) and is presented as percentage.
Time Frame: Period 3: Week 24, 15 minutes pre-dose (Period was 24 weeks)
Population: Safety Analysis Set included all participants who received at least one dose of study drug in the considered period. Number analyzed = participants evaluable for the endpoint at the specified timepoints. As pre-specified, data were collected and are reported pooled for all dose levels in Period 3 and are presented at the specified timepoint.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Period 3: Encaleret
Number analyzed (Participants) | 13
percentage | 0.016 (0.004)

10. Secondary Outcome: Periods 1, 2 and 3: Urinary Calcium Clearance as Assessed by 24-Hour Total Excretion
Time Frame: Periods 1 and 2: Day 5; Period 3, Week 24 (Period was 5 days for Periods 1 and 2; 24 weeks for Period 3)
Population: Safety Analysis Set, which included all participants who received at least one dose of study drug in the considered period. Number analyzed = participants evaluable for the endpoint at the specified timepoints. As pre-specified, data were collected and are reported pooled for all dose levels in Period 2 and Period 3 at the specified timepoints. As pre-specified, data were collected and are presented per dose at the specified timepoint for Period 1.
Measure: Mean (Standard Deviation); unit: mg/24hr
Arm/Group | Period 1: Encaleret | Period 2: Encaleret | Period 3: Encaleret
Number analyzed (Participants) | 3 | 13 | 13
mg/24hr
  Period 1: Day 5 AM 180 mg; PM 180 mg: number analyzed (Participants) | 3 | 0 | 0
  Period 1: Day 5 AM 180 mg; PM 180 mg | 84 (146) |  |
  Period 1: Day 5 AM 180 mg; PM 120 mg: number analyzed (Participants) | 1 | 0 | 0
  Period 1: Day 5 AM 180 mg; PM 120 mg | 0 (NA) — Standard deviation could not be calculated as there was only 1 participant with evaluable data. |  |
  Period 2: Day 5: number analyzed (Participants) | 0 | 13 | 0
  Period 2: Day 5 |  | 179 (108) |
  Period 3: Week 24: number analyzed (Participants) | 0 | 0 | 13
  Period 3: Week 24 |  |  | 202 (83)

11. Secondary Outcome: Periods 1, 2 and 3: Renal Function as Assessed by Estimated Glomerular Filtration Rate (eGFR)
Description: eGFR was calculated using Chronic Kidney Disease - Epidemiology Collaboration (CKD-EPI) formula (mL/min/1.73m^2) = 141 x min (SCr/K, 1)^α x max(SCR /K,1)-1.209 x 0.993Age x 1.018 [if female] x 1.159 [if Black], where SCr is the serum creatinine (mg/dL), K = 0.7 for female and 0.9 for males, α is -0.329 for female and -0.411 for males.
Time Frame: Periods 1 and 2: Day 5 (15 minutes pre-dose), Period 3: Week 24 (15 minutes pre-dose) (Period was 5 days for Periods 1 and 2; 24 weeks for Period 3)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Period 1: Encaleret | Period 2: Encaleret | Period 3: Encaleret
Number analyzed (Participants) | 6 | 13 | 13
mL/min/1.73m^2
  Period 1: Day 5 AM (180 mg): number analyzed (Participants) | 6 | 0 | 0
  Period 1: Day 5 AM (180 mg) | 91.1 (18.73) |  |
  Period 2: Day 5 AM: number analyzed (Participants) | 0 | 13 | 0
  Period 2: Day 5 AM |  | 90.6 (25.30) |
  Period 3: Week 24: number analyzed (Participants) | 0 | 0 | 13
  Period 3: Week 24 |  |  | 82.0 (21.10)

12. Secondary Outcome: Periods 1, 2 and 3: Serum Levels of 1,25-(OH)2 Vitamin D
Time Frame: Periods 1 and 2: Day 5 (15 minutes pre-dose), Period 3: Week 24 (15 minutes pre-dose); (Period was 5 days for Periods 1 and 2; 24 weeks for Period 3)
Population: Safety Analysis Set, all participants who received at least 1 dose of study drug in the considered period. Overall number of participants analyzed=participants evaluable for the endpoint. Number analyzed=participants evaluable for the endpoint at specified timepoints. As pre-specified, data were collected and reported pooled for all dose levels in Period 2 and 3 at the specified timepoints. As pre-specified, data were collected and are reported per dose at the specified timepoint for Period 1.
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/mL)
Arm/Group | Period 1: Encaleret | Period 2: Encaleret | Period 3: Encaleret
Number analyzed (Participants) | 6 | 13 | 13
picograms per milliliter (pg/mL)
  Period 1: Day 5 AM (180 mg): number analyzed (Participants) | 6 | 0 | 0
  Period 1: Day 5 AM (180 mg) | 25.8 (12.24) |  |
  Period 2: Day 5 AM: number analyzed (Participants) | 0 | 13 | 0
  Period 2: Day 5 AM |  | 30.5 (16.40) |
  Period 3: Week 24: number analyzed (Participants) | 0 | 0 | 13
  Period 3: Week 24 |  |  | 31.2 (16.19)

13. Secondary Outcome: Periods 1, 2 and 3: Magnesium, Phosphorus, and Creatinine Levels as Assessed by Blood Sample Examinations
Time Frame: as for outcome 12
Population: Safety Analysis Set, all participants who received at least one dose of study drug in the considered period. Overall number of participants analyzed=participants evaluable for the endpoint. Number analyzed=participants evaluable for the endpoint at specified timepoints. As pre-specified, data were collected and reported pooled for all dose levels in Period 2 and 3 at specified timepoints. As pre-specified, data were collected and are presented per dose at the specified timepoint for Period 1.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Period 1: Encaleret | Period 2: Encaleret | Period 3: Encaleret
Number analyzed (Participants) | 6 | 13 | 13
mg/dL
  ⦁ Magnesium - Period 1: Day 5 AM (180 mg): number analyzed (Participants) | 6 | 0 | 0
  ⦁ Magnesium - Period 1: Day 5 AM (180 mg) | 2.2 (0.36) |  |
  Magnesium - Period 2: Day 5 AM: number analyzed (Participants) | 0 | 13 | 0
  Magnesium - Period 2: Day 5 AM |  | 1.9 (0.28) |
  Magnesium - Period 3: Week 24: number analyzed (Participants) | 0 | 0 | 13
  Magnesium - Period 3: Week 24 |  |  | 2.0 (0.20)
  ⦁ Phosphorus - Period 1: Day 5 AM (180 mg): number analyzed (Participants) | 6 | 0 | 0
  ⦁ Phosphorus - Period 1: Day 5 AM (180 mg) | 2.9 (0.39) |  |
  Phosphorus - Period 2: Day 5 AM: number analyzed (Participants) | 0 | 13 | 0
  Phosphorus - Period 2: Day 5 AM |  | 3.1 (0.75) |
  Phosphorus - Period 3: Week 24: number analyzed (Participants) | 0 | 0 | 13
  Phosphorus - Period 3: Week 24 |  |  | 3.7 (0.52)
  ⦁ Creatinine - Period 1: Day 5 AM (180 mg): number analyzed (Participants) | 6 | 0 | 0
  ⦁ Creatinine - Period 1: Day 5 AM (180 mg) | 0.93 (0.188) |  |
  Creatinine - Period 2: Day 5 AM: number analyzed (Participants) | 0 | 13 | 0
  Creatinine - Period 2: Day 5 AM |  | 0.94 (0.229) |
  Creatinine - Period 3: Week 24: number analyzed (Participants) | 0 | 0 | 13
  Creatinine - Period 3: Week 24 |  |  | 1.01 (0.212)

14. Secondary Outcome: Periods 1, 2 and 3: Creatinine, Phosphorus, Magnesium, and Citrate Total Excretion Levels as Assessed by Urine Sample Examinations
Time Frame: Periods 1 and 2: Day 5 (0-24h post-dose), Period 3: Week 24 (0-24h post-dose); (Period was 5 days for Periods 1 and 2; 24 weeks for Period 3)
Population: Safety Analysis Set, all participants who received at least one dose of study drug in the considered period. Overall number of participants analyzed=participants evaluable for the endpoint. Number analyzed=participants evaluable for the endpoint at the specified timepoints. As pre-specified, data were collected and reported pooled for all dose levels in Period 2 and 3 at specified timepoints. As pre-specified, data were collected and are reported per dose at the specified timepoint for Period 1.
Measure: Mean (Standard Deviation); unit: mg/24hr
Arm/Group | Period 1: Encaleret | Period 2: Encaleret | Period 3: Encaleret
Number analyzed (Participants) | 3 | 13 | 13
mg/24hr
  Creatinine - Period 1: Day 5 AM 180 mg, PM 180 mg: number analyzed (Participants) | 3 | 0 | 0
  Creatinine - Period 1: Day 5 AM 180 mg, PM 180 mg | 1454 (248) |  |
  Creatinine - Period 1: Day 5 AM 180 mg, PM 120 mg: number analyzed (Participants) | 1 | 0 | 0
  Creatinine - Period 1: Day 5 AM 180 mg, PM 120 mg | 1190 (NA) — Standard deviation could not be calculated as there was only 1 participant with evaluable data. |  |
  Creatinine - Period 2: Day 5: number analyzed (Participants) | 0 | 13 | 0
  Creatinine - Period 2: Day 5 |  | 1408 (367) |
  Creatinine - Period 3: Week 24: number analyzed (Participants) | 0 | 0 | 13
  Creatinine - Period 3: Week 24 |  |  | 1345 (373)
  Phosphorus - Period 1: Day 5 AM 180 mg, PM 180 mg: number analyzed (Participants) | 3 | 0 | 0
  Phosphorus - Period 1: Day 5 AM 180 mg, PM 180 mg | 877 (353) |  |
  Phosphorus - Period 1: Day 5 AM 180 mg, PM 120 mg: number analyzed (Participants) | 1 | 0 | 0
  Phosphorus - Period 1: Day 5 AM 180 mg, PM 120 mg | 1100 (NA) — Standard deviation could not be calculated as there was only 1 participant with evaluable data. |  |
  Phosphorus - Period 2: Day 5: number analyzed (Participants) | 0 | 13 | 0
  Phosphorus - Period 2: Day 5 |  | 962 (226) |
  Phosphorus - Period 3: Week 24: number analyzed (Participants) | 0 | 0 | 13
  Phosphorus - Period 3: Week 24 |  |  | 754 (240)
  Magnesium - Period 1: Day 5 AM 180 mg, PM 180 mg: number analyzed (Participants) | 3 | 0 | 0
  Magnesium - Period 1: Day 5 AM 180 mg, PM 180 mg | 104 (5) |  |
  Magnesium - Period 1: Day 5 AM 180 mg, PM 120 mg: number analyzed (Participants) | 1 | 0 | 0
  Magnesium - Period 1: Day 5 AM 180 mg, PM 120 mg | 110 (NA) — Standard deviation could not be calculated as there was only 1 participant with evaluable data. |  |
  Magnesium - Period 2: Day 5: number analyzed (Participants) | 0 | 13 | 0
  Magnesium - Period 2: Day 5 |  | 161 (66) |
  Magnesium - Period 3: Week 24: number analyzed (Participants) | 0 | 0 | 13
  Magnesium - Period 3: Week 24 |  |  | 121 (38)
  Citrate - Period 1: Day 5 AM 180 mg, PM 180 mg: number analyzed (Participants) | 3 | 0 | 0
  Citrate - Period 1: Day 5 AM 180 mg, PM 180 mg | 662 (77) |  |
  Citrate - Period 1: Day 5 AM 180 mg, PM 120 mg: number analyzed (Participants) | 1 | 0 | 0
  Citrate - Period 1: Day 5 AM 180 mg, PM 120 mg | 778 (NA) — Standard deviation could not be calculated as there was only 1 participant with evaluable data. |  |
  Citrate - Period 2: Day 5: number analyzed (Participants) | 0 | 13 | 0
  Citrate - Period 2: Day 5 |  | 381 (203) |
  Citrate - Period 3: Week 24: number analyzed (Participants) | 0 | 0 | 12
  Citrate - Period 3: Week 24 |  |  | 439 (224)

15. Secondary Outcome: Periods 1, 2 and 3: pH as Assessed by Urine Sample Examinations
Time Frame: Periods 1 and 2: Day 5 (0-24 hours post-dose), Period 3: Week 24: (0-24 hours post-dose); (Period was 5 days for Periods 1 and 2; 24 weeks for Period 3)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Period 1: Encaleret | Period 2: Encaleret | Period 3: Encaleret
Number analyzed (Participants) | 3 | 13 | 11
pH
  Period 1: Day 5 AM 180 mg; PM 180 mg 0-24 hours post-dose: number analyzed (Participants) | 3 | 0 | 0
  Period 1: Day 5 AM 180 mg; PM 180 mg 0-24 hours post-dose | 6.2 (2.02) |  |
  Period 1: Day 5 AM 180 mg; PM 120 mg 0-24 hours post-dose: number analyzed (Participants) | 1 | 0 | 0
  Period 1: Day 5 AM 180 mg; PM 120 mg 0-24 hours post-dose | 5.0 (NA) — Standard deviation could not be calculated as there was only one participant with evaluable data. |  |
  Period 2: Day 5 0-24 hours post-dose: number analyzed (Participants) | 0 | 13 | 0
  Period 2: Day 5 0-24 hours post-dose |  | 6.1 (0.68) |
  Period 3: Week 24 0-24 hours post-dose: number analyzed (Participants) | 0 | 0 | 11
  Period 3: Week 24 0-24 hours post-dose |  |  | 6.5 (0.69)

16. Secondary Outcome: Periods 1, 2 and 3: Potassium and Sodium Total Excretion Levels as Assessed by Urine Sample Examinations
Time Frame: as for outcome 14
Population: Safety Analysis Set, all participants who received at least one dose of study drug in the considered period. Overall number of participants analyzed=participants evaluable for the endpoint. Number analyzed=participants evaluable for the endpoint at specified timepoints. As pre-specified, data were collected and reported pooled for all dose levels in Period 2 and 3 at specified timepoints. As pre-specified, data were collected and are reported per dose at the specified timepoint for Period 1.
Measure: Mean (Standard Deviation); unit: Milliequivalents (meq)/24hr
Arm/Group | Period 1: Encaleret | Period 2: Encaleret | Period 3: Encaleret
Number analyzed (Participants) | 3 | 13 | 13
Milliequivalents (meq)/24hr
  Potassium Period 1: Day 5 AM 180 mg, PM 180 mg: number analyzed (Participants) | 3 | 0 | 0
  Potassium Period 1: Day 5 AM 180 mg, PM 180 mg | 79.00 (48.662) |  |
  Potassium Period 1: Day 5 AM 180 mg, PM 120 mg: number analyzed (Participants) | 1 | 0 | 0
  Potassium Period 1: Day 5 AM 180 mg, PM 120 mg | 82.00 (NA) — Standard deviation could not be calculated as there was only one participant with evaluable data. |  |
  Potassium Period 2: Day 5: number analyzed (Participants) | 0 | 13 | 0
  Potassium Period 2: Day 5 |  | 69.38 (24.476) |
  Potassium Period 3: Week 24: number analyzed (Participants) | 0 | 0 | 13
  Potassium Period 3: Week 24 |  |  | 61.46 (32.196)
  Sodium Period 1: Day 5 AM 180 mg, PM 180 mg: number analyzed (Participants) | 3 | 0 | 0
  Sodium Period 1: Day 5 AM 180 mg, PM 180 mg | 186.33 (84.831) |  |
  Sodium Period 1: Day 5 AM 180 mg, PM 120 mg: number analyzed (Participants) | 1 | 0 | 0
  Sodium Period 1: Day 5 AM 180 mg, PM 120 mg | 192.00 (NA) — Standard deviation could not be calculated as there was only one participant with evaluable data. |  |
  Sodium Period 2: Day 5: number analyzed (Participants) | 0 | 13 | 0
  Sodium Period 2: Day 5 |  | 184.77 (51.038) |
  Sodium Period 3: Week 24: number analyzed (Participants) | 0 | 0 | 13
  Sodium Period 3: Week 24 |  |  | 182.23 (95.407)

17. Secondary Outcome: Periods 1, 2 and 3: Cyclic Adenosine Monophosphate (cAMP) Total Excretion Levels as Assessed by Urine Sample Examinations
Time Frame: Periods 1 and 2: Day 5 (0-4h post-dose), Period 3: Week 24 (0-4h post dose); (Period was 5 days for Periods 1 and 2; 24 weeks for Period 3)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: nanomoles per deciliter (nmol/dL)
Arm/Group | Period 1: Encaleret | Period 2: Encaleret | Period 3: Encaleret
Number analyzed (Participants) | 5 | 13 | 11
nanomoles per deciliter (nmol/dL)
  Period 1: Day 5 AM, 180 mg, PM 180 mg, 0-4 hours post-dose: number analyzed (Participants) | 5 | 0 | 0
  Period 1: Day 5 AM, 180 mg, PM 180 mg, 0-4 hours post-dose | 2.98 (0.795) |  |
  Period 1: Day 5, AM 180 mg, PM 120 mg 0-4 hours post-dose: number analyzed (Participants) | 1 | 0 | 0
  Period 1: Day 5, AM 180 mg, PM 120 mg 0-4 hours post-dose | 2.90 (NA) — Standard deviation could not be calculated as there was only one participant with evaluable data. |  |
  Period 2: Day 5 0-4 hours post-dose: number analyzed (Participants) | 0 | 13 | 0
  Period 2: Day 5 0-4 hours post-dose |  | 2.79 (0.762) |
  Period 3: Week 24 0-4 hours post-dose: number analyzed (Participants) | 0 | 0 | 11
  Period 3: Week 24 0-4 hours post-dose |  |  | 2.68 (0.704)

18. Secondary Outcome: Periods 1, 2 and 3: Bone Resorption Markers as Assessed by Collagen Cross-Linked C-Telopeptide (CTx)
Description: Blood samples were taken for analysis of bone resorption markers (CTx).
Time Frame: Periods 1 and 2: Day 5 (15 minutes pre-dose), Period 3 Week 24 (15 minutes pre-dose); (Period was 5 days for Periods 1 and 2; 24 weeks for Period 3)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Picograms per milliliter (pg/mL)
Arm/Group | Period 1: Encaleret | Period 2: Encaleret | Period 3: Encaleret
Number analyzed (Participants) | 6 | 13 | 13
Picograms per milliliter (pg/mL)
  Period 1: Day 5 AM 180 mg: number analyzed (Participants) | 6 | 0 | 0
  Period 1: Day 5 AM 180 mg | 386 (165) |  |
  Period 2: Day 5 AM: number analyzed (Participants) | 0 | 13 | 0
  Period 2: Day 5 AM |  | 266 (161) |
  Period 3: Week 24: number analyzed (Participants) | 0 | 0 | 13
  Period 3: Week 24 |  |  | 744 (565)

19. Secondary Outcome: Periods 1, 2 and 3: Bone Formation Markers as Assessed by Blood Procollagen Type 1 N-Propeptide (P1NP)
Description: Blood samples were taken for analysis of bone formation markers (P1NP).
Time Frame: as for outcome 18
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Micrograms per liter (mcg/L)
Arm/Group | Period 1: Encaleret | Period 2: Encaleret | Period 3: Encaleret
Number analyzed (Participants) | 6 | 13 | 13
Micrograms per liter (mcg/L)
  Period 1: Day 5 AM 180 mg: number analyzed (Participants) | 6 | 0 | 0
  Period 1: Day 5 AM 180 mg | 27.33 (5.007) |  |
  Period 2: Day 5 AM: number analyzed (Participants) | 0 | 13 | 0
  Period 2: Day 5 AM |  | 26.8 (12.25) |
  Period 3: Week 24: number analyzed (Participants) | 0 | 0 | 13
  Period 3: Week 24 |  |  | 103.7 (87.20)

ADVERSE EVENTS:
Time Frame: Up to 16 months
Description: All-cause mortality is reported for all enrolled participants. Serious and other adverse events are reported for the Safety Analysis Set, which included all participants who received at least one dose of study drug in the considered period. As pre-specified in the protocol, data were collected and are presented pooled for Periods 2 and 3. As pre-specified, data were collected and are presented pooled for all cohorts and doses for Period 1 and for Periods 2 and 3 combined.
Arm/Group | Period 1: Encaleret | Periods 2 and 3: Encaleret
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/13
Other Adverse Events (participants affected / at risk) | 5/6 | 13/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Period 1: Encaleret (N=6) | Periods 2 and 3: Encaleret (N=13)
Upper respiratory tract infection (Infections and infestations) | 0 | 4
Vulvovaginal mycotic infection (Infections and infestations) | 0/3 | 3/8 — Number at risk adjusted as this is a sex-specific event.
Pharyngitis (Infections and infestations) | 1 | 1
Bacterial vaginosis (Infections and infestations) | 0/3 | 1/8 — Number at risk adjusted as this is a sex-specific event.
Chronic sinusitis (Infections and infestations) | 0 | 1
Green nail syndrome (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 9
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 6
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 5
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Heat exhaustion (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 4
Constipation (Gastrointestinal disorders) | 0 | 3
Dizziness (Nervous system disorders) | 0 | 3
Headache (Nervous system disorders) | 1 | 2
Paraesthesia (Nervous system disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 2
Injection site reaction (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Blood pressure decreased (Investigations) | 1 | 1
Weight decreased (Investigations) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 2
Superficial vein thrombosis (Vascular disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hypocitraturia (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-05-18): https://cdn.clinicaltrials.gov/large-docs/29/NCT04581629/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-26): https://cdn.clinicaltrials.gov/large-docs/29/NCT04581629/SAP_001.pdf